CLINICAL TRIAL: NCT04034875
Title: SOCIALBI, a Rasch Questionnaire for the Evaluation of Anger, Hostility and Aggression After Acquired Brain Injury.
Brief Title: Questionnaire for the Evaluation of Anger, Hostility and Aggression After Acquired Brain Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of clinical trial unit, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-SOCIALBI
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Lesion
Keywords: Acquired cerebral lesion; Anger; Aggression
MeSH Terms: conditions — Aggression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with acquired brain injury (Experimental)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — questionnaire

SUMMARY:
The incidence of aggression and violent behavior is usually reported to be high after acquired brain injury, around 54%. Behaviors with verbal agression and, less frequently, physical agressions, are described.

These behaviors may be linked to the dysfunction of the frontal lobes responsible for executive functions and complex social interactions, or to the dysfunction of the temporal structures that may also be responsible for increased aggression.

It is interesting to note that very few scales or specific questionnaires evaluate the factors and co-variables that could lead to aggressive behavior after an acquired brain injury. Such questionnaires are very rare, and none have been validated in French.

The objective of this study is to develop a questionnaire in French that aims to assess anger, hostility and aggression after acquired brain injury. The psychometric qualities of this questionnaire will be evaluated using the Rasch probabilistic model.

The development of such a tool will be of major interest for clinical practice and future clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the CHU Brugmann Hospital
* Central neurological pathology of vascular or traumatic origin, acute or chronic (known since more than one year).

Exclusion Criteria:

* Pregnant or lactating women
* Presence or antecedents of psychiatric disease
* Degenerative pathology (ex: Parkinson...)
* Antecedents of other neurologic pathologies before the acquired lesion
* Oral or written comprehension dysfunctions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Questionnaire evaluation by Rasch methodology | 30 minutes
  questionnaire validity

CONTACTS AND LOCATIONS:
Overall Officials: Eric Durand, MD, Principal Investigator — CHU Brugmann
Locations (3):
- Brugmann University Hospital, Brussels, Belgium
- France (2):
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Hôpitaux Saint Maurice, Saint-Maurice

IPD SHARING:
Plan to Share IPD: No